CLINICAL TRIAL: NCT04067427
Title: To Reduce Recurrence of Symptomatic Atrial Fibrillation and Improve Quality of Life After Catheter Ablation for Atrial Fibrillation by App-based Mental Training (Mental AF)
Brief Title: Reducing Recurrence of Symptomatic Atrial Fibrillation After Catheter Ablation by App-based Mental Training
Acronym: Mental-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Health Institute GmbH (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAF2019
Record Dates: First submitted 2019-08-15; First posted 2019-08-26 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Meditation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental training (Active Comparator): AF ablation followed by 3 months of a daily app-based mental training for 10 to 15 minutes per session. AF 6 questionnaire will be answered weekly via the Mental-AF webpage.
  Interventions: Other: Mental training
- Control (No Intervention): AF ablation without subsequent mental training. AF 6 questionnaire will be answered weekly via the Mental-AF webpage.

INTERVENTIONS:
Other: Mental training — App-based mental training
  Arms: Mental training

SUMMARY:
Atrial fibrillation (AF) is one of the most common heart rhythm disorders and it is associated with a variety of symptoms leading to a considerable deterioration in quality of life. The Mental-AF trial is intended to inquire if an app-based mental training can reduce the occurrence of symptomatic AF episodes within the blanking period, i.e. the first three months after catheter ablation for AF.

DETAILED DESCRIPTION:
To explore the potential of a daily app-based mindfulness mental training in improving AF symptoms, assessed by self-reported outcome measures, i.e. the AF 6 questionnaire, AF Effect on QualiTy of Life (AFEQT) and Patient Reported Outcome Measurement Information System (PROMIS) Global Health questionnaires, as well as in reducing AF burden in 7-day-Holter, within the first 12 weeks following AF ablation.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing AF ablation with symptomatic paroxysmal or chronic atrial fibrillation (EHRA II-IV)
* Availability of smart phone with the capability to run android 5 or iOS 9 or newer versions
* Capability to use mobile phone applications
* Internet access
* Consent to study participation

Exclusion Criteria:

* Patients < 18 years of age
* Unavailability of smart phone running at least Android 5 or iOS 9
* Pregnancy

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation (AF) 6 questionnaire score | 12 weeks, assessed weekly
  Atrial fibrillation specific symptomatic outcome defined by AF 6 sum scores during the first 12 weeks following AF ablation, based on a 10-point Likert scale, ranging from 0 (no symptoms) to 10 (severe symptoms), sum scores ranging from 0 to 60.

SECONDARY OUTCOMES:
Atrial Fibrillation Effect on QualiTy of Life (AFEQT) score | Follow up (3 months)
  Effects of AF on quality of Life, assessed by a 20-item questionnaire with 4 conceptual domains (daily Activities, treatment concern, symptoms and treatment satisfaction) on a 7-point Likert scale, responses ranging from 1 (no symptoms/limitations) to 7 (most severe limitations/symptoms), higher scores indicating better health status, the raw scores can be transformed to a 0 to 100 scale adjusting for missing data
Patient-Reported Outcome Measurement Information System (PROMIS) Global Health 10 score | Follow up (3 months)
  PROMIS Global Health questionnaire for the assessment of physical and mental health domains by 10 items using a 5-point Likert scale, ranging from (5) excellent to (1) poor. Higher scores indicate a healthier patient.
Atrial fibrillation burden | Follow up (3 months)
  Time in AF as assessed in 7-day-Holter
Heart Rate | Follow up (3 months)
  Heart Rate during blood pressure measurement
Blood pressure | Follow up (3 months)
  Office blood pressure measurement of diastolic and systolic blood pressure
Atrial Fibrillation Effect on QualiTy of Life (AFEQT) score | Follow up at 12 months
  Effects of AF on quality of Life, assessed by a 20-item questionnaire with 4 conceptual domains (daily Activities, treatment concern, symptoms and treatment satisfaction) on a 7-point Likert scale, responses ranging from 1 (no symptoms/limitations) to 7 (most severe limitations/symptoms), higher scores indicating better health status, the raw scores can be transformed to a 0 to 100 scale adjusting for missing data

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Lurz, Principal Investigator — Herzzentrum Leipzig, Strümpellstr. 39, 04289 Leipzig, Germany
Locations (1):
- Leipzig Heart Institute, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lurz J, Hengelhaupt L, Unterhuber M, Stenzel L, Hilbert S, Schober AR, Dinov B, Darma A, Dagres N, Hindricks G, Lurz P, Bollmann A. App-Based Mental Training to Reduce Atrial Fibrillation-Related Symptoms After Pulmonary Vein Isolation: MENTAL AF Trial. J Am Heart Assoc. 2024 Jun 4;13(11):e033500. doi: 10.1161/JAHA.123.033500. Epub 2024 May 23. PMID 38780185